CLINICAL TRIAL: NCT02757326
Title: A Phase Ib/II Safety and Efficacy Study of ABC294640 in Patients With Refractory or Relapsed Multiple Myeloma Who Have Previously Been Treated With Proteasome Inhibitors and Immunomodulatory Drugs
Brief Title: ABC294640 (Opaganib) in Refractory / Relapsed Multiple Myeloma
Acronym: ABC-103
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Expiration of National Cancer Institute (NCI) funding of the study.
Sponsor: RedHill Biopharma Limited (Industry)
Collaborators: Apogee Biotechnology Corporation (Industry); Duke University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00062304; 1R44CA199767-01 (NIH)
Record Dates: First submitted 2016-03-31; First posted 2016-05-02 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma
Keywords: sphingosine kinase 2 inhibitor; sphingosine kinase 2; SK2 inhibitor; SK2
MeSH Terms: conditions — Multiple Myeloma | interventions — 3-(4-chlorophenyl)-adamantane-1-carboxylic acid (pyridin-4-ylmethyl)amide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase Ib/II (Experimental): For Phase Ib, the planned ABC294640 (Opaganib) doses for the escalation phase are: 250, 500, and 750 mg BID given continuously. The dose will be given under fasting conditions (at least 1 hour before or 2 hours after eating). One cycle is 28 days of treatment.
  For phase II study, the patients will be treated with single agent ABC294640 at the MTD determined from the phase IB study (or at the highest dose used, if MTD is not reached) until disease progression or intolerable toxicity occurs in an individual patient.
  Interventions: Drug: Opaganib

INTERVENTIONS:
Drug: Opaganib — Opaganib, [3-(4-chlorophenyl)-adamantane-1-carboxylic acid (N-(Pyridin-4-ylmethyl)pyridine-4-carboxamide) amide, hydrochloride salt] is an orally available inhibitor of the enzyme SK2.
  Other Names: ABC294640

SUMMARY:
This is a Phase Ib/II safety and efficacy trial of single agent ABC294640, an inhibitor of sphingosine kinase 2 and dihydroceramide desaturase, in refractory or relapsed multiple myeloma (MM). Cohorts of patients with refractory or relapsed MM who have previously been treated with proteasome inhibitors and immunomodulatory agents will receive increasing doses of oral ABC294640. The starting dosage for ABC294640 will be 250 mg bis in die (BID) which is known to be safely tolerated as a single agent, and the ABC294640 dose will be escalated to two additional dose cohorts of 500 and 750 mg BID using Bayesian model average continual reassessment method (BMA-CRM) for dose finding. It is expected that 18 patients will be used to determine the maximum tolerated dose (MTD) for ABC294640 in refractory or relapsed MM. Up to 56 additional patients will be treated on the phase II portion of the study at the MTD or maximum dose used in phase I, with interim stopping rules for futility.

Pharmacokinetic (PK) and pharmacodynamic (PD) assessments of ABC294640 will be conducted on Day 1 of Cycle 1. Bone marrow biopsy will be obtained prior to the initiation of ABC294640, at the end of cycle #3 and at the end of cycle #6. In addition to serum protein electrophoresis (SPEP), urine protein electrophoresis (UPEP) and serum free light chain measurement, correlative studies will be performed to measure sphingosine kinase 2 (SK2) activity, sphingosine metabolites, and additional biomarkers in CD138+ myeloma cells.

DETAILED DESCRIPTION:
Objectives for Phase 1b:

Primary Objectives • To assess safety and determine the maximum tolerated dose (MTD) of single agent ABC294640 in patients with refractory or relapsed multiple myeloma (MM) who have been previously treated with proteasome inhibitors and immunomodulatory agents.

Secondary Objectives

* To assess the antitumor activity of single agent ABC294640 in patients with refractory or relapsed MM after 3 cycles of treatment.
* To determine the pharmacokinetics of ABC294640 following administration of the drug.
* To describe the effects of ABC294640 on plasma levels of sphingosine 1-phosphate and IL-6 (interleukin - 6) in patients with refractory or relapsed MM.
* To assess pharmacodynamic markers (SK2 mRNA (messenger ribonucleic acid) level or activity, sphingolipid metabolites, c-Myc, Mcl-1 and pS6) in bone marrow CD138+ myeloma cells.

Objectives for Phase 2:

Primary Objectives

• Assess overall treatment response rate and overall survival in patients with relapsed or refractory MM treated with single-agent ABC294640.

Secondary Objectives

* To assess the treatment response of ABC294640 in patients with refractory or relapsed MM after 3 cycles of treatment.
* To determine if pharmacodynamic markers (SK2 mRNA or activity, sphingolipid metabolites, c-Myc, Mcl-1 and pS6) in bone marrow CD138+ myeloma cells predict tumor response to the treatment with ABC294640.

The projected ABC294640 doses for the escalation phase are: 250, 500, and 750 mg BID orally continuously as determined in the single agent trial for ABC294640. The dose will be given under fasting conditions (at least 1 hour before or 2 hours after eating). Each cycle of treatment is 28 days.

Patients will be monitored for safety and pharmacodynamics effects weekly in Cycle 1, biweekly for Cycles 2-4, and monthly for subsequent cycles.

Myeloma treatment response will be assessed as follows:

* Serum protein electrophoresis (SPEP), urine protein electrophoresis (UPEP) and serum free light chains before each cycle.
* Skeletal survey at screening, then every year or at the end of study if the study ends before the anniversary.
* Bone marrow biopsy and aspirates at the last day of cycle #3 and cycle #6 (± 7 days).

For the phase II portion of the study, patients will be treated with single agent ABC294640 at the MTD determined from the phase Ib study (or highest dose used, if MTD is not reached) until disease progression or intolerable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a diagnosis of symptomatic multiple myeloma, relapsed or refractory after previous treatment with a proteasome inhibitor (bortezomib or carfilzomib) and an immunomodulatory agent (thalidomide, lenalidomide or pomalidomide).
2. Have measurable disease as defined by at least one of the following:

   * Serum monoclonal (M) protein ≥1.0 g/dl by protein electrophoresis
   * >200 mg of M protein in the urine on 24 hour electrophoresis
   * Serum immunoglobulin free light chain ≥10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
   * Monoclonal bone marrow plasmacytosis ≥30%
3. Voluntary signed and dated institutional review board (IRB) approved informed consent form in accordance with regulatory and institutional guidelines.
4. Time interval from last systemic chemotherapy (not including low dose dexamethasone) more than 2 weeks prior to initiation of ABC294640. Patients receiving high dose dexamethasone defined as 40mg dexamethasone a day for 4 days will need 2 weeks washout prior to initiation of ABC294640
5. 18 years of age or older.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
7. Acceptable liver function:

   * Bilirubin ≤ 1.5 times upper limit of normal (CTCAE Grade 1 baseline)
   * AST (aminotransferase) (SGOT), ALT (alanine aminotransferase) (SGPT) ≤ 5 x ULN (CTCAE Grade 2 baseline)
   * Serum creatinine ≤1.5 XULN (1.5 times the upper limit of normal) (CTCAE Grade 1 baseline)
8. Acceptable hematologic status (with or without transfusion support):

   * Absolute neutrophil count ≥1000 cells/mm3,
   * Platelet count ≥50,000 (plt/mm3),
   * Hemoglobin ≥9 g/dL.
9. Urinalysis: No clinically significant abnormalities.
10. PT (partial thromboplastin) and PTT (partial thromboplastin time) ≤ 1.5 X ULN after correction of nutritional deficiencies that may contribute to prolonged PT/PTT.
11. As determined by the treating investigator, the patient must have well-controlled blood pressure, defined as systolic blood pressure <150mmHg (Millimeter of Mercury)and/or diastolic blood pressure <100 mmHg for the majority of measurements.
12. A negative pregnancy test (if female of child bearing potential).
13. For men and women of child-producing potential, willingness to use effective contraceptive methods during the study.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Patients who are currently participating in any other clinical trial of an investigational product.
3. Major surgery within 30 days prior to start of treatment
4. Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to start of treatment
5. Known human immunodeficiency virus infection
6. Active hepatitis B or C infection with abnormal liver functions (i.e., LFTs (liver function test) > 2 x upper normal limits)
7. Unstable angina or myocardial infarction within 4 months prior to start of treatment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker
8. Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to start of treatment
9. Nonhematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder
10. Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to initiation of ABC294640
11. Any other clinically significant medical or psychiatric disease or condition, or social situation that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yubin Kang, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venkata JK, An N, Stuart R, Costa LJ, Cai H, Coker W, Song JH, Gibbs K, Matson T, Garrett-Mayer E, Wan Z, Ogretmen B, Smith C, Kang Y. Inhibition of sphingosine kinase 2 downregulates the expression of c-Myc and Mcl-1 and induces apoptosis in multiple myeloma. Blood. 2014 Sep 18;124(12):1915-25. doi: 10.1182/blood-2014-03-559385. PMID 25122609
- [Derived] Kang Y, Sundaramoorthy P, Gasparetto C, Feinberg D, Fan S, Long G, Sellars E, Garrett A, Tuchman SA, Reeves BN, Li Z, Liu B, Ogretmen B, Maines L, Ben-Yair VK, Smith C, Plasse T. Phase I study of opaganib, an oral sphingosine kinase 2-specific inhibitor, in relapsed and/or refractory multiple myeloma. Ann Hematol. 2023 Feb;102(2):369-383. doi: 10.1007/s00277-022-05056-7. Epub 2022 Dec 3. PMID 36460794

RESULTS

PARTICIPANT FLOW:
Groups:
- 250 mg: Unblinded Phase 1b dose-finding study with dose escalation of study drug ABC294640 (Opaganib). Once a subject was determined to be eligible for the study, the subject was enrolled in the dose escalation Phase 1b study testing ABC294640 at 250 mg twice a day (bis in die). A cycle of treatment was defined as 28 days and doses were given initially under fasting conditions. Subsequent to a food effect study, treatment was given after a light to moderate meal.
- 500 mg: Unblinded Phase 1b dose-finding study with dose escalation of study drug ABC294640. Once a subject was determined to be eligible for the study, the subject was enrolled in the dose escalation Phase 1b study testing ABC294640 at 500 mg twice a day). A cycle of treatment was defined as 28 days and doses were given initially under fasting conditions. Subsequent to a food effect study, treatment was given after a light to moderate meal.
- 750 mg: Unblinded Phase 1b dose-finding study with dose escalation of study drug ABC294640. Once a subject was determined to be eligible for the study, the subject was enrolled in the dose escalation Phase 1b study testing ABC294640 doses at 750 mg twice a day ). A cycle of treatment was defined as 28 days and doses were given initially under fasting conditions. Subsequent to a food effect study, treatment was given after a light to moderate meal.
Period: Overall Study
Arm/Group | 250 mg | 500 mg | 750 mg
Started | 3 | 4 | 6
Completed | 3 | 4 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with Refractory or Relapsed Multiple Myeloma Who have Previously Been Treated with Proteasome Inhibitors and Immunomodulatory Agents were treated with three doses of ABC294640.
Groups:
- Phase 1b - 250 mg BID: For Phase 1b, ABC294640 was dosed at 250 BID given continuously. The dose was given under fasting conditions (at least 1 hour before or 2 hours after eating). One cycle is 28 days of treatment.
- Phase 1b - 500 mg BID: For Phase 1b, ABC294640 was dosed at 500 BID given continuously. The dose was given under fasting conditions (at least 1 hour before or 2 hours after eating). One cycle is 28 days of treatment
- Phase 1b - 750 mg BID: For Phase 1b, ABC294640 was dosed at 750 mg BID given continuously. The dose was given under fasting conditions (at least 1 hour before or 2 hours after eating). One cycle is 28 days of treatment
- Total: Total of all reporting groups
Arm/Group | Phase 1b - 250 mg BID | Phase 1b - 500 mg BID | Phase 1b - 750 mg BID | Total
Number analyzed (Participants) | 3 | 4 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (4.58) | 75.8 (13.94) | 63.8 (6.94) | 68.9 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 1 | 6
  Male | 2 | 0 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 3 | 6
  White | 3 | 1 | 3 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 6 | 13
Baseline ECOG (Eastern Cooperative Oncology Group)Status [Count of Participants; unit: Participants] — Lower ECOG grades correlate with a better clinical status:
  Grade 0- Fully active, able to carry on all pre-disease performance without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. -Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours
  3. -Capable of only limited self-care, confined to a bed or chair >50% of waking hours
  4. - Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  5. - Dead
  Participants
    ECOG 0 | 0 | 0 | 1 | 1
    ECOG 1 | 2 | 4 | 3 | 9
    ECOG 2 | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: Evaluation of three doses of opaganib - 250 mg bid, 500 mg bid and 750 mg bid to determine the maximum tolerated dose (MTD) based upon the dose limiting toxicity (DLT) using a Bayesian model averaging continual reassessment method and is the dose at which the estimated probability of toxicity is closest to the target probability 0.33 among all doses.
Time Frame: 6 months
Population: Safety population
Measure: Number; unit: mg
Groups:
- Opaganib: Unblinded Phase 1b dose-finding study with dose escalation of study drug ABC294640. Once a subject was determined to be eligible for the study, the subject was enrolled in the dose escalation Phase 1b study testing ABC294640 at 250, 500 and 750 mg twice a day. A cycle of treatment was defined as 28 days and doses were given initially under fasting conditions. Subsequent to a food effect study, treatment was given after a light to moderate meal.
Arm/Group | Opaganib
Number analyzed (Participants) | 13
mg | NA — The maximum tolerated dose was not reached in the study

2. Secondary Outcome: To Assess the Antitumor Activity of Single Agent Opaganib in Patients With Refractory or Relapsed Multiple Myeloma After 3 Cycles of Treatment.
Description: Stable disease, partial response, complete response or disease progression.
Time Frame: After 3 cycles (12 weeks) of treatment
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Groups:
- ABC294640 250 mg BID; ABC294640 500 mg BID: ABC294640 250 mg BID given continuously
- ABC294640 750 mg BID: ABC294640 750 mg BID given continuously
Arm/Group | ABC294640 250 mg BID | ABC294640 500 mg BID | ABC294640 750 mg BID
Number analyzed (Participants) | 3 | 4 | 6
Participants | 0 | 2 | 0

3. Secondary Outcome: Number of Patients With Dose Limiting Toxicity
Description: For the phase 1b portion of the trial, a dose-limiting toxicity (DLT) was defined as an adverse event at least possibly related to the study medication:
  Non-hematologic DLT is defined as any Grade 3 or greater ADR (adverse drug reaction), except symptomatic AEs such as nausea, vomiting, and diarrhea which could be reduced to less than Grade 3 within 72 hours with standard supportive measures (i.e., antiemetics and antidiarrheals).
  Hematologic DLT is defined as
  * Grade 4 neutropenia or thrombocytopenia that lasts more than 7 days after the last dose of study drug
  * or greater than or equal to Grade 3 thrombocytopenia in the presence of greater than or equal to Grade 3 hemorrhage of any organ/site
  * or any Grade 5 hematologic toxicity
Time Frame: 12 months
Population: All participants receiving any amount of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ABC294640 250 mg BID | ABC294640 500 mg BID | ABC294640 750 mg BID
Number analyzed (Participants) | 3 | 4 | 6
Participants | 0 | 0 | 1

4. Secondary Outcome: Maximum Concentration (Cmax) of ABC294640
Description: To determine the Cmax of ABC294640 following administration of the drug.
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: mcg/hr/mL
Groups:
- ABC294640 250 mg BID; ABC294640 500 mg BID; ABC294640 750 mg BID: Samples for PK were drawn on Day 1 of Cycle 1 immediately before dosing and at 1, 2, 4, and 8 hours after dosing.
Arm/Group | ABC294640 250 mg BID | ABC294640 500 mg BID | ABC294640 750 mg BID
Number analyzed (Participants) | 3 | 4 | 6
mcg/hr/mL | 5.6 (1.7) | 12.5 (2.5) | 25.8 (3)

ADVERSE EVENTS:
Time Frame: Up to 20.5 weeks
Description: Treatment emergent adverse events (TEAE) were any event not present before exposure to study medication or any event already present that worsens in either intensity or frequency following exposure to study drug.
Groups:
- 250 mg Phase 1b: For Phase 1b, ABC294640 was dosed at 250 BID given continuously. The dose was given under fasting conditions (at least 1 hour before or 2 hours after eating). One cycle is 28 days of treatment.
- 500 mg Phase 1b: For Phase 1b, ABC294640 was dosed at 500 BID given continuously. The dose was given under fasting conditions (at least 1 hour before or 2 hours after eating). One cycle is 28 days of treatment.
- 750 mg Phase 1b: For Phase 1b, ABC294640 was dosed at 750 BID given continuously. The dose was given under fasting conditions (at least 1 hour before or 2 hours after eating). One cycle is 28 days of treatment.
Arm/Group | 250 mg Phase 1b | 500 mg Phase 1b | 750 mg Phase 1b
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/4 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 250 mg Phase 1b (N=3) | 500 mg Phase 1b (N=4) | 750 mg Phase 1b (N=6)
ALTERED MENTAL STATUS (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) — 250 mg cohort, Grade 3, NOT RELATED
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) — Grade 3, Not related, Drug interrupted
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Grade 2, not related, dose not changed
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Colitis- not related to therapy
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Worsening constipation not related to therapy
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Hip fracture not related to therapy - Grade 3
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Cardiac arrest not related to therapy - Grade 4
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Impending pathological fracture, right femur, not therapy related - Grade 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 250 mg Phase 1b (N=3) | 500 mg Phase 1b (N=4) | 750 mg Phase 1b (N=6)
Summary of Adverse events occurring in >10% of patients by System Organ Class and Preferred Term (Blood and lymphatic system disorders) | 3 (28) | 4 (34) | 6 (41)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 3 (3) | 3 (3)
Lymphocyte count decreased (Investigations) | 3 (3) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
International normalized ratio (Investigations) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight (Investigations) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT02757326/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT02757326/SAP_001.pdf
  • Informed Consent Form (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT02757326/ICF_002.pdf